CLINICAL TRIAL: NCT06763991
Title: Safety and Efficacy of Connecting the Residual Ear to the Cartilage Scaffold in First- vs. Second-Stage Surgery : a Protocl of a Randomized Controlled Trial in Non-expanded Auricular Reconstruction for Concha-type Microtia
Brief Title: Safety and Efficacy of Connecting the Residual Ear to the Cartilage Scaffold in First- vs. Second-Stage Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sichuan Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Xinjie Zhang, Principal investigator, Sichuan Provincial People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-256-1
Record Dates: First submitted 2025-01-03; First posted 2025-01-08 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Microtia; Outcome Assessment; RCT; Surgery Related Complications Rate; Treatment Outcome; Reconstruction
MeSH Terms: conditions — Congenital Microtia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- First-stage Connection (Active Comparator): After obtaining written informed consent, eligible patients will be randomized with a 1:1 allocation using an online randomization module. A random number will be assigned sequentially to make sure that every patient will be randomly allocated into two groups (Accepting First-stage Connection and Second-stage Connection).
  Interventions: Procedure: One-stage connection
- Two-stage connection (Experimental): After obtaining written informed consent, eligible patients will be randomized with a 1:1 allocation using an online randomization module. A random number will be assigned sequentially to make sure that every patient will be randomly allocated into two groups (Accepting One-stage connection and Two-stage connection).
  Interventions: Procedure: Two-stage connection

INTERVENTIONS:
Procedure: Two-stage connection — Two-stage connection refers to a procedure that connecting and incorporating the cartilage framework with the residual ear during the second stage surgery of ear reconstruction. An intact cartilage framework is embedded in skin pocket in the first stage, hence, in the second stage of surgery, parts of the cartilage framework that has already survived will be shaved off to ensure the firm combination between the residual era cartilage and grafted costal cartilage.
  Arms: Two-stage connection
Procedure: One-stage connection — One-stage connection refers to a procedure that connecting and incorporating the cartilage framework with the residual ear in the first stage surgery of ear reconstruction. In one-stage surgery, the cartilage framework is connected with the residual ear (non-deformed, unexcluded part) to form a smooth and complete ear subunit structure. In this way, it is necessary to trim the excess postauricular skin, which may pose a greater risk of blood supply. After the first stage of surgery, the overall appearance of surgical ear is already roughly similar to that of a normal ear.
  Arms: First-stage Connection

SUMMARY:
Eligible patients will be admitted from the outpatient clinic to complete the relevant examinations after admission（Preoperative routine examination and chest CT）. The baseline parameters will be registered when admitted to hospital, including case number, diagnosis, sex, age, height, weight, and underlying medical conditions. Patients have at least 12 hours to consider participation in the study and will be given the opportunity to ask questions about the study. Written informed consent will be obtained by the surgical resident or the surgeon after admission to the hospital.

Randomization will be done by relevant member . After inclusion, patients will be allocated to one of the two study groups (First-stage Connection or Second-stage Connection) using an online randomization program. The perioperative care will be the same for all included patients.Surgery will be performed by experienced surgeons, with non-expanded ear reconstruction using autologous rib cartilage. The surgery normally comprises two stages. After each surgery, details and duration of the surgery will be documented. For each stage of surgery, patients are scheduled for visits about 3-6 months. In addition, after the total surgery, patients are to fill out 'Glasgow Benefit Inventory' and 'Patient and Observer Scar Assessment Scale'.

ELIGIBILITY:
Inclusion Criteria:

All consecutive patients between 6 and 30 years with a congenital concha-microtia8, admitted to our hospital are potentially eligible, and enrollment in the study will be based on the following criteria.

1. Patients were fully informed about the purpose, modalities and risks associated with this study, signed an informed consent form and were willing to be followed up.
2. Contrast-enhanced computed tomography (CT) scan shows he or she has 3.Patients can tolerate general anesthesia without severe chronic organic or mental illness.

Exclusion Criteria:

1. Patients combined with other ear diseases such as ear fistula, titis media, etc.
2. Patients receive other unrelated ear surgeries during the study
3. Skin in the surgical area with infection, ulceration, and scarring.

Ages: 6 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 78 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2027-02-20 (Estimated); Study Completion 2027-02-20 (Estimated)

PRIMARY OUTCOMES:
Grade-A healing | For each stage of surgery, patients are scheduled for visits about 3-6 months.
  Grade-A healing is defined as optimal wound alignment, epidermal integrity, and tight subcutaneous tissue junctions, with no significant inflammatory response or complications during recovery, and the stitches can be removed within 10 days after the operation.

SECONDARY OUTCOMES:
complication rates | For each stage of surgery, patients are scheduled for visits about 3-6 months.
  Incidence of infection, hematoma, flap necrosis, skin necrosis, and cartilage scaffold exposure
Scar score | 3-6 months after the total ear reconstruction surgery
  The Patient and Observer Scar Assessment Scale (POSAS) is a validated and applicable tool for scar evaluation. There are two numeric scales of POSAS, one for patients and another for observers. Each of items receives a score from 1 to 10. A score of 1 represents normal skin and 10 represents the worst scar imaginable. To add the scores of each item, a total score of the observer scale ranges from 5 to 50, and a patient scale ranges from 6 to 60. The lowest scores, 5 and 6, respectively, reflect normal skin. The higher the scores, the worse the scar.
Patients' satisfaction score | 3-6 months after the total ear reconstruction surgery
  To evaluate patients' satisfaction of the final result after surgery, we use Glasgow benefit inventory(GBI) as a evaluated tool. GBI comprises 18 items. Each item is scored using the Likert 5-level scoring scale. The GBI total score can range from -100 (maximum adverse effect) through 0 (no effect) to 100 (maximum benefit). In addition, subscores can be calculated: a general subscore, a social support score and a physical health score.

CONTACTS AND LOCATIONS:
Locations (1):
- Sichuan provincial people's hospital, Chengdu, Sichuan, China

REFERENCES:
- [Derived] Zhang X, Chen Z, Chen M, Wang Y, Du L, Cai Z, Jiang Z. Safety and efficacy of connecting the residual ear to the cartilage scaffold in the first-stage versus second-stage surgery: a protocol of a randomised controlled trial in non-expanded auricular reconstruction for concha-type microtia. BMJ Open. 2026 Feb 4;16(2):e104106. doi: 10.1136/bmjopen-2025-104106. PMID 41638738